CLINICAL TRIAL: NCT02416583
Title: Concurrent Oxytocin With Membrane Sweeping Versus Dinoprostone Pessary in Labor Induction of Nulliparas at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyo Hoon Park, MD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWP_PG_N2
Record Dates: First submitted 2015-04-01; First posted 2015-04-15 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Failed Induction of Labor
Keywords: membrane sweeping; dinoprostone; nulliparas; labor induction
MeSH Terms: interventions — Oxytocin; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin & Membrane sweeping (Active Comparator): Women assigned to "Concurrent oxytocin with membrane sweeping" had their cervix swept by inserting the examining finger as high as possible past the internal cervical os, followed by oxytocin infusion the next day
  Interventions: Drug: Oxytocin; Procedure: Membrane sweeping
- Oxytocin & Dinoprostone (Active Comparator): For women assigned to "Concurrent oxytocin with dinoprostone vaginal insert": The 10mg dinoprostone vaginal insert were placed in the posterior fornix for cervical ripening, followed by oxytocin infusion the next day
  Interventions: Drug: Oxytocin; Drug: Dinoprostone

INTERVENTIONS:
Drug: Oxytocin
Drug: Dinoprostone
  Arms: Oxytocin & Dinoprostone
Procedure: Membrane sweeping
  Arms: Oxytocin & Membrane sweeping

SUMMARY:
To compare concurrent oxytocin with membrane sweeping versus dinoprostone pessary in labor induction for nulliparas at term with an unfavorable cervix

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* Nulliparous women
* gestational age >=37.0 weeks
* Bishop score <=6
* intact amniotic membrane
* absence of labor
* live fetus with vertex presentation
* no previous uterine surgical procedure

Exclusion Criteria:

* Multiple pregnancy
* Placenta previa

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery within 24 hours | From the time of initiating intervention (i.e.concurrent membrane sweeping with dinoprostone or only dinoprostone) until the time of vaginal delivery, assessed up to 24 hours
  Vaginal delivery within 24 hours is defined as vaginal delivery after 24 hours of initiating intervention (i.e.concurrent membrane sweeping with dinoprostone or only dinoprostone) on the first day of induction.

SECONDARY OUTCOMES:
Successful labor induction | From the time of initiating intervention (i.e.concurrent membrane sweeping with dinoprostone or only dinoprostone) until the time of active phase of labor ( defined as a cervical dilatation of >=4cm), assessed up to 24 hours
  to achieve the active phase of labor corresponding to a cervical dilatation of >=4cm
Incidence of cesarean delivery | End of labor induction (assessed up to 120 hours)
  From the time of initiating intervention (i.e.concurrent membrane sweeping with dinoprostone or only dinoprostone) until the time of cesarean delivery, assessed up to 120 hours
The interval from start of oxytocin to delivery | From the time of initiating oxytocin infusion until the time of delivery, assessed up to 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea